CLINICAL TRIAL: NCT05155163
Title: Stepped Care for Patients to Optimize Whole Recovery
Acronym: SC-POWR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000031094; 1RM1DA055310-01 (NIH)
Record Dates: First submitted 2021-12-07; First posted 2021-12-13 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Opioid Use Disorder; Chronic Pain
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment as Usual (No Intervention): Treatment as usual for opioid use disorder
- SC-POWR (Experimental): Treatment as usual for opioid use disorder with the addition of CBT with possible stepped care to exercise and stress reduction
  Interventions: Behavioral: SC-POWR

INTERVENTIONS:
Behavioral: SC-POWR — Patients assigned to SC-POWR receive 12 Cognitive Behavioral Therapy (CBT) sessions over 24 weeks.
  Arms: SC-POWR

SUMMARY:
This is a prospective, randomized clinical trial of 204 patients with opioid use disorder (OUD) and chronic pain (CP) to test the effectiveness of treatment as usual compared with Stepped Care for Patients to Optimize Whole Recovery (SC-POWR) to reduce pain interference (Aim 1) and decrease illicit opioid use, alcohol use, anxiety, depression, and stress, and improve sleep (Aim 2). Eligible participants will begin medications for opioid use disorder (MOUD) and will be randomized to receive SC-POWR (i.e., cognitive behavioral therapy (CBT), MOUD, and onsite groups for exercise [Wii Fit, Tai Chi] and stress reduction [relaxation training, auricular acupuncture] for 24 weeks. Participants will be followed for another 24 weeks to evaluate durability of treatment response on pain interference illicit opioid use, alcohol use, anxiety, depression, stress, sleep, and retention in MOUD (Aim 3).

DETAILED DESCRIPTION:
Participants who meet criteria for CP and OUD (N=204) will be initiated onto MOUD and randomized to 24 weeks of either treatment as usual (TAU) or 24 weeks of SC-POWR. SC-POWR patients will be "stepped up" according to a priori criteria. Patients randomized to SC-POWR will receive a behavioral intervention consisting of 12 Cognitive Behavioral Therapy (CBT) sessions over a 24-week period involving improvements in substance use and pain since baseline. Following 24 weeks of SC-POWR, patients are offered once monthly peer-support groups.

This study receives support from and included in the HEAL Initiative (https://heal.nih.gov/).

ELIGIBILITY:
Inclusion Criteria:

* Seeking treatment at APT Foundation
* Receiving medications for opioid use disorder (MOUD provided by APT)
* Have high impact chronic pain (>= 3 months duration of pain occurring most days which limits life or work activities and/or leads to inability to work)
* Meet DSM-5 criteria for moderate to severe OUD
* In the past 2 months, has an opioid-positive urine test or self-reports opioid use
* Understand English
* Able to provide informed consent

Exclusion Criteria:

* Have pending surgery or invasive pain management procedure
* Acutely psychotic, suicidal, or homicidal
* Psychiatric instability (e.g., recent suicide attempt)
* Have a contraindication to exercise (e.g. complete heart block)
* Have a pending or planned relocation or pending incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain interference using The Pain, Enjoyment of Life and General Activity (PEG) Scale | Baseline, weekly for 24 weeks, weeks 36 and 48
  Pain interference is measured using the PEG scale, a 3-item scale with each item scored from 0-10. Total scores are achieved by averaging the 3 items. Total sore range from 0-10. Higher scores indicate more pain and interference.

SECONDARY OUTCOMES:
Change in alcohol use | Baseline, weekly for 24 weeks, weeks 36 and 48
  Measured by the TLFB. The Timeline Followback for alcohol uses a calendar to record amount of alcohol consumed over a desired time period.
Change in Anxiety symptoms using General Anxiety Disorder-7 (GAD-7) | Baseline, weekly for 24 weeks, weeks 36 and 48
  General Anxiety Disorder- 7 (GAD-7) is a 7 item self report instrument that measures anxiety Items are scored on a 4-point scale, ranging from "not at all (0)" to "nearly everyday (3)". Item scores are summed with a total score ranging from 0 to 21: 0-4 Minimal anxiety; 5-9 Mild anxiety; 10-14 Moderate anxiety; 15-21 Severe anxiety.
Change in Depression assessed using Patient Health Questionnaire-9 (PHQ-9) | Baseline, monthly for 24 weeks, weeks 36 and 48
  PHQ-9 assesses depression symptoms. Each item asks about the frequency of specific depressive symptoms experienced over the past two weeks. The response options are scored from 0 to 3, indicating "not at all" to "nearly every day." The total score on the PHQ-9 ranges from 0 to 27, with higher scores indicating greater severity of depressive symptoms. The scoring can also be divided into categories, with scores of 0-4 indicating minimal or no depression, 5-9 indicating mild depression, 10-14 indicating moderate depression, 15-19 indicating moderately severe depression, and 20 or above indicating severe depression.
Change in pain intensity assessed using the Brief Pain Inventory (BPI) | Baseline, weekly for 24 weeks, weeks 36 and 48
  The BPI has a total score range of 0-10 where: 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-10 = severe pain. Total pain severity score can be found by averaging all items.
Change in sleep | Baseline, weekly for 24 weeks, weeks 36 and 48
  Measured by a single sleep item from the Brief Pain Inventory (BPI). Higher scores mean greater pain interference with sleep.
Change in stress assessed using the Perceived Stress Scale (PSS) | Baseline, monthly for 24 weeks, weeks 36 and 48
  The PSS is a 10-item self- report scale. PSS scores are obtained by reversing responses to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. Total score range from 0-40 with higher scores indicate greater levels of stress.
Change in composite illicit opioid use | Baseline, weekly for 24 weeks, weeks 36 and 48
  Opioid use is measured by the Timeline Followback (TLFB) and confirmed by urine drug testing. The TLFB uses a calendar to measure opioid or other drug use over a desired time period; it is a self-reported measure of drug use. To confirm the self report, a urine test will be performed to detect the presence of opioids.

CONTACTS AND LOCATIONS:
Overall Officials: Declan Barry, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - APT Foundation, New Haven, Connecticut
  - APT Foundation, North Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No